CLINICAL TRIAL: NCT01130155
Title: IMPACT2: Monitoring Interventions to Improve ACT Access and Targeting
Brief Title: IMPACT2: Monitoring Interventions to Improve Artemisinin-based Combination Therapy (ACT) Access and Targeting
Acronym: IMPACT2
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: London School of Hygiene and Tropical Medicine (Other)
Collaborators: Ifakara Health Institute (Other); Centers for Disease Control and Prevention (U.S. Federal Agency); Bill and Melinda Gates Foundation (Other)
Responsible Party: Catherine Goodman, LSHTM
Other Study IDs: PHGBVG04
Record Dates: First submitted 2010-05-24; First posted 2010-05-25 (Estimated); Last update posted 2011-06-23 (Estimated); Status verified 2011-06

CONDITIONS: Malaria; Anaemia
Keywords: Antimalarials; Diagnosis; Access to treatment; Quality of care
MeSH Terms: conditions — Malaria; Anemia; Disease

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- Mwanza Region: Households, and patients presenting at public health facilities in Mwanza Region
- Mbeya Region: Households, and patients presenting at public health facilities in Mbeya Region
- Mtwara Region: Households, and patients presenting at public health facilities in Mtwara Region

SUMMARY:
It is generally agreed that artemisinin-based combination therapy (ACT) is the malaria therapy of choice but there is much less agreement about the best ACT-deployment strategies. Countries are now beginning to adopt policies to enhance ACT deployment that aim to address 2 key goals: (i) making ACTs more readily and speedily accessible to patients: or (ii) targeting ACTs to patients shown to have malaria parasitaemia.

The Tanzanian Government has secured funding to address both ACT access and targeting on a national scale. Access is to be improved through the distribution of subsidised ACTs through private facilities and retail drug shops under the Affordable Medicines Facility-malaria (AMFm). Targeting is to be addressed through enhancing microscopy and introducing rapid diagnostic tests (RDTs) in health facilities at every level of the system.

This study will evaluate these two interventions in 3 rural regions of Tanzania which are all expected to receive both interventions during the study period. The investigators will assess the effectiveness of the interventions in terms of coverage, equity, quality, adherence, and public health impact using a pre-post plausibility design based on before and after household, health facility and outlet surveys. The null hypothesis is that the interventions will have no impact on the coverage of prompt effective treatment for fever and malarial. In addition, the investigators will estimate the cost and cost-effectiveness of implementation from a health system and household perspective. Finally the investigators will explore the socio-cultural context and other factors that influence the implementation and outcome of the interventions.

ELIGIBILITY:
Inclusion Criteria:

* Household survey - All consenting and assenting residents available in selected households
* Health facility survey - patients presenting to selected health facilities with fever or history of fever in the prior 24 hours; Age >= 3 months, or Weight ≥ 5 kg; First visit to this health facility for this illness episode

Exclusion Criteria:

* Household survey - Children less than 3 months of age will be excluded from providing a blood sample
* Health facility survey - Signs of severe illness

Min Age: 3 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: For the household survey, all selected households in Mtwara, and Mwanza and Mbeya Regions in Tanzania.
  For the health facility survey patients presenting to selected health facilities with fever or history of fever in the prior 24 hours.
Sampling Method: Probability Sample
Enrollment: 33900 (Estimated)
Dates: Start 2010-05; Primary Completion 2012-09 (Estimated); Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
Percent of population reporting fever in last two weeks that received ACT within 24hrs/48hrs
Percent of population reporting fever in last two weeks that got a finger/heel stick for a malaria diagnostic test within 24hrs/48hrs
Proportion of patients presenting to public health facilities with fever who receive a diagnostic test for malaria
Proportion of patients presenting to public health facilities with fever who receive rapid diagnostic test (RDT) for malaria and are appropriately treated according to RDT results

SECONDARY OUTCOMES:
Percent of patients receiving an ACT that adhered to full dose with correct dose timing
Mean and median household cost per febrile episode
The accuracy of RDTs performed by health workers
Adequacy of health facility resources for diagnosis and treatment of malaria

CONTACTS AND LOCATIONS:
Overall Officials: Catherine Goodman, PhD, Principal Investigator — London School of Hygiene and Tropical Medicine; Patrick Kachur, MD, Principal Investigator — Centers for Disease Control and Prevention; Salim Abdulla, PhD, Principal Investigator — Ifakara Health Institute
Locations (1):
- Ifakara Health Institute, Dar es Salaam, Tanzania